CLINICAL TRIAL: NCT04854486
Title: Impact of GSE and Xylitol (Xlear) in Symptoms and Time to PCR Negativisation of Patients With Acute COVID-19 Infection
Brief Title: Impact of GSE and Xylitol (Xlear) on COVID-19 Symptoms and Time to PCR Negativisation in COVID-19 Patients
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Study Period Ended / Not Completed
Sponsor: Larkin Community Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: LCH-2-112020
Record Dates: First submitted 2021-04-17; First posted 2021-04-22 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Covid19
Keywords: intranasal spray; Covid19
MeSH Terms: conditions — COVID-19 | interventions — Xylitol

STUDY DESIGN:
Intervention Model Description: Placebo controlled
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Treatment Group (Experimental): Xylitol + GSE
  Interventions: Other: GSE and Xylitol
- Control placebo (Placebo Comparator): Saline
  Interventions: Drug: Control Placebo

INTERVENTIONS:
Other: GSE and Xylitol — Participants are given the experimental treatment to be used for 7 days.
  Arms: Treatment Group
Drug: Control Placebo — Saline
  Arms: Control placebo

SUMMARY:
This clinical trial aims to ascertain the impact of GSE and Xylitol (XLEAR) in decreasing the time of negativisation in PCR testing in patients with COVID-19.

ELIGIBILITY:
Inclusion Criteria

* Adults of ages 18 to 90 years of both sexes
* With positive SARS-CoV-2 carriage confirmed by nasopharyngeal PCR
* Signed informed consent
* 1- Mild symptoms: Minimum respiratory symptoms or asymptomatic plus positive test
* 2- Moderate symptoms: Respiratory symptoms such as cough, mild shortness of breath with mild oxygen desaturation(room air SpO2 <92% and >88% or <88% corrected to >92% with 2lt of oxygen)

Exclusion Criteria

* Patients with Severe symptoms: Hypoxia (SpO2 <88% not corrected by 2 lt nc oxygen) plus severe shortness of breath (excluded)
* Patient with very low viral load (threshold cycle [Ct] > 25 per PCR).
* Known hypersensitivity to one of the constituents, particularly to xylitol or GSE
* Under 18 years of age
* Women of childbearing age who are pregnant, breastfeeding mothers, and intend to become pregnant during the study period; unwilling/unable to take a pregnancy test.
* Unable to provide informed consent or decline to consent or unwillingness to adhere to the Standard of Care protocol.
* Patients with severe symptoms -Hypoxia (SpO2 <88% not corrected by 2 liter non- concentrated oxygen) plus severe shortness of breath
* History of immunodeficiency or are currently receiving immunosuppressive therapy.
* Have had a planned surgical procedure within the past 12 weeks.
* Already part of this trial, recruited at a different hospital.
* Patient unable to perform oro-nasopharyngeal decolonization
* Patients with acute exacerbation of severe comorbidities like heart disorders Chronic Obstructive Pulmonary Disease (COPD), Heart Failure New York Heart Association (NYHA) Class 3 and 4 and/or diseases with severe oxygenation problems
* Patients on Remdesivir and/or other clinical trials.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2021-12-16 (Actual); Primary Completion 2022-03-30 (Actual); Study Completion 2022-11-16 (Actual)

PRIMARY OUTCOMES:
Change of time to negativisation via PCR | Baseline and 7 days
  There will be a change in the time to negativisation via PCR as compared to the average 14-day time to negative result.

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - Larkin Community Hospital Palm Springs Campus, Miami, Florida
  - Larkin Community Hospital, Miami, Florida

IPD SHARING:
Plan to Share IPD: No